CLINICAL TRIAL: NCT04220255
Title: Clinical Outcome at 5 Years After Implantation of Medicontur Multifocal Intraocular Lens Liberty 677MY: Visual Outcomes, Patients' Satisfaction, YAG Capsulotomy Rate
Brief Title: Clinical Outcome at 5 Years After Implantation of the Liberty677MY Multifocal Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MC_Liberty677MY_HU_2019
Record Dates: First submitted 2019-12-20; First posted 2020-01-07 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Liberty677MY Multifocal IOL — multifocal intraocular lens (IOL)

SUMMARY:
The study will assess visual outcomes, light disturbances and patients' satisfaction after implantation with the Liberty677MY multifocal IOL, as well as protection of PCO development within 5 year follow-up.

DETAILED DESCRIPTION:
The Liberty677MY multifocal IOL is designed for restoring near, intermediate and distance vision. The technology of Liberty 677MY is based on the elevated phase shift technology (patent pending). Previous evaluations showed the strength of studied IOL both in laboratory and clinical conditions.

Patients will be examined 5 years after implantation. The examination will include the measurement of the best corrected distance, intermediate and near visual acuity (assessed with Early Treatment Diabetic Retinopathy Study (ETDRS) charts), intraocular pressure (contact Goldman tonometry), biomicroscopic and fundocsopic examination, contrast sensitivity (CSV-1000), defocus curve, reading capability, pupilometry in different light conditions and PCO evaluation, Nd:YAG capsulotomy rate, photo-documentation of anterior segment. YAG capsulotomy will be indicated in case of posterior capsule opacification (PCO). The criteria for YAG capsulotomy will be visual acuity decreased 2 or more lines when using (ETDRS) charts. Details of all related and unrelated complications will be documented, including severity, time of onset, specific treatment and clinical outcome. The investigators will also record whether the capsulorhexis is on or partially off the optic.

ELIGIBILITY:
Inclusion Criteria:

* pseudophakic patients implanted with Liberty 677MY in 2014-2015 during the study under the ethical approval: 059823/2014/OTIG

Exclusion Criteria:

* diabetic retinopathy
* iris neovascularisation
* serious intraoperative complications
* congenital eye abnormality
* glaucoma
* pseudoexfoliation syndrome
* amblyopia
* uveitis
* long-term anti-inflammatory treatment
* AMD (advanced AMD)
* retinal detachment
* prior ocular surgery in personal medical history (except cataract surgery aiming the implantation of the multifocal IOL)
* previous laser treatment
* corneal diseases
* severe retinal diseases (dystrophy, degeneration)
* severe myopia (if required IOL power is lower than 10 D)
* inadequate visualization of the fundus on preoperative examination
* patients deemed by the clinical investigator because of any systemic disease.
* pregnancy
* eye trauma in medical history
* current use of systemic steroids or topical ocular medication
* preoperative smaller pupil size of 6 mm under topical mydriasis
* kappa angle >5°

Ages: 40 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pseudophakic patients implanted with Liberty 677MY in 2014-2015 during the study under the ethical approval: 059823/2014/OTIG
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Uncorrected Decimal VA (6 m) | 5 years after implantation
  Visual acuity (VA) was tested monocularly (each eye separately) and binocularly (both eyes together) 5 years after implantation, unaided at a distance of 6 meters (m) using Early Treatment Diabetic Retinopathy ( ETDRS) charts and assessed in logarithm of the minimum angle of resolution (LogMAR).
Uncorrected Decimal VA (60 cm) | 5 years after implantation
  Visual acuity (VA) was tested monocularly (each eye separately) and binocularly (both eyes together) 5 years after implantation, unaided at a distance of 60 centimeters (cm) using ETDRS charts, assessed in LogMAR.
Uncorrected Decimal VA (40 cm) | 5 years after implantation
  Visual acuity (VA) was tested monocularly (each eye separately) and binocularly (both eyes together) 5 years after implantation, unaided at a distance of 40 centimeters (cm) using ETDRS charts, assessed in LogMAR.
Corrected Decimal VA (6 m) | 5 years after implantation
  Visual acuity (VA) was tested monocularly (each eye separately) and binocularly (both eyes together) 5 years after implantation, unaided at a distance of 6 meters (m) using ETDRS charts, assessed in LogMAR.
Corrected Decimal VA (60 cm) | 5 years after implantation
  Visual acuity (VA) was tested monocularly (each eye separately) and binocularly (both eyes together) 5 years after implantation, unaided at a distance of 60 centimeters (cm) using ETDRS charts , assessed in LogMAR.
Corrected Decimal VA (40 cm) | 5 years after implantation
  Visual acuity (VA) was tested monocularly (each eye separately) and binocularly (both eyes together) 5 years after implantation, unaided at a distance of 40 centimeters (cm) using ETDRS charts, assessed in LogMAR.
Defocus Curve Profiles | 5 years after implantation
  Visual acuity measurement (assessed in logarithm of the minimum angle of resolution (LogMAR)) taken with different levels of optical defocus was tested monocularly (each eye separately) and binocularly (both eyes together).
Contrast Sensitivity CSV-1000 | 5 years after implantation
  Binocular Assessment of contrast sensitivity at threshold using the Contrast sensitivity vision (CSV) CSV-1000 in photopic and mesopic conditions with or without glare.

SECONDARY OUTCOMES:
Posterior capsule opacification (PCO) rate | 5 years after implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Retinaszervíz Kft, Veszprém, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gyory JF, Srinivasan S, Madar E, Balla L. Long-term performance of a diffractive-refractive trifocal IOL with centralized diffractive rings: 5-year prospective clinical trial. J Cataract Refract Surg. 2021 Oct 1;47(10):1258-1264. doi: 10.1097/j.jcrs.0000000000000670. PMID 33974369